CLINICAL TRIAL: NCT05334121
Title: Randomized Clinical Trial to Analyze the Safety of Chronic Intake of a β-alanine Supplement in Active Individuals
Brief Title: Safety Analysis of Chronic Intake of a β-alanine Supplement
Acronym: HIPOX-β
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UCAMCFE-00025
Record Dates: First submitted 2022-03-26; First posted 2022-04-19 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-03

CONDITIONS: Product Safety
MeSH Terms: interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product - Beta Alanine (Experimental): The product will be consumed every day for 4 weeks. Four intakes of 3g each, separated by three hours each, will be carried out.
  Interventions: Dietary Supplement: Beta-alanine
- Control group - Placebo (Placebo Comparator): The product will be consumed every day for 4 weeks. Four intakes of 3g each, separated by three hours each, will be carried out.
  Interventions: Other: Control product consumption

INTERVENTIONS:
Dietary Supplement: Beta-alanine — The product will be consumed every day for 4 weeks. Four intakes of 3g each, separated by three hours each, will be carried out.
  Arms: Product - Beta Alanine
Other: Control product consumption — Product with identical characteristics to the experimental product. The product will be consumed every day for 4 weeks. Four intakes of 3g each, separated by three hours each, will be carried out.
  Arms: Control group - Placebo

SUMMARY:
Single-center, double-blind, placebo-controlled clinical trial with two arms (product and placebo) to analyze the safety of beta-alanine consumption in active people.

DETAILED DESCRIPTION:
After recruitment, subjects will be randomized and assigned to one of the two arms of the study: beta-alanine group or control group (placebo).

Subjects must be active people, and will take a dose of 15 g per day of the product for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 40 years of age.
* Physically active people. They must train at least 3 sessions per week.
* Have been training continuously for at least one year.

Exclusion Criteria:

* Participant suffering from chronic illness.
* Serious or terminal illness.
* Suffering from a lasting injury that prevents him/her from training in the month prior to the intervention.
* Inability to understand the informed consent.
* Previous experience in the consumption of beta alanine.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Liver safety variables | Change in hepatic safety after 8 weeks of consumption
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

SECONDARY OUTCOMES:
Paresthesia test | Change after 8 weeks of consumption
  Visual analogue scale (1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Fco Javier López Román, Principal Investigator — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain

REFERENCES:
- [Derived] Maestre-Hernandez AB, Perez-Pinero S, Lopez-Roman FJ, Andreu-Caravaca L, Luque-Rubia AJ, Ramos-Campo DJ, Diaz-Silvestre MJ, Avila-Gandia V. Effect of a sustained-release formulation of beta-alanine on laboratory parameters and paresthesia in recreational trained men: a randomized double-blind placebo-controlled study. Front Nutr. 2023 Sep 12;10:1213105. doi: 10.3389/fnut.2023.1213105. eCollection 2023. PMID 37766731